CLINICAL TRIAL: NCT03922945
Title: A Phase IV, Multi-Center, Randomized, Double-Blind, Placebo-Controlled, Parallel-Design Study to Determine the Safety and Efficacy of VI-0521 in Obese Adolescents
Brief Title: A Phase IV Safety and Efficacy Study of VI-0521 in Adolescents With Obesity
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: VIVUS LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OB-403
Record Dates: First submitted 2019-04-16; First posted 2019-04-22 (Actual); Results first posted 2022-09-10 (Actual); Last update posted 2022-09-10 (Actual); Status verified 2022-08

CONDITIONS: Adolescent Obesity; Obesity in Adolescence; Adolescent Overweight
Keywords: weight loss; obesity; weight control
MeSH Terms: conditions — Pediatric Obesity; Weight Loss; Obesity | interventions — Qsymia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- VI-0521 Mid Dose (Phentermine 7.5 mg +Topiramate 46 mg) (Experimental): Weeks 1-2: VI-0521 (Phentermine 3.75 mg + Topiramate 23 mg) oral capsule, once daily; Weeks 3-56: VI-0521 (Phentermine 7.5 mg + Topiramate 46 mg) oral capsule, once daily
  Interventions: Drug: VI-0521 oral capsule; Behavioral: Lifestyle Modification
- VI-0521 Top Dose (Phentermine 15 mg + Topiramate 92 mg) (Experimental): Weeks 1-2: VI-0521 (Phentermine 3.75 mg + Topiramate 23 mg) oral capsule, once daily; Weeks 3-12: VI-0521 (Phentermine 7.5 mg + Topiramate 46 mg) oral capsule, once daily; Weeks 13-14: VI-0521 (Phentermine 11.25 mg + Topiramate 69 mg) oral capsule, once daily; Weeks 15-56: VI-0521 (Phentermine 15 mg + Topiramate 92 mg) oral capsule, once daily
  Interventions: Drug: VI-0521 oral capsule; Behavioral: Lifestyle Modification
- Placebo (Placebo Comparator): Subjects will receive placebo oral capsule, once daily for up to 56 weeks
  Interventions: Drug: Placebo oral capsule; Behavioral: Lifestyle Modification

INTERVENTIONS:
Drug: VI-0521 oral capsule — Phentermine/Topiramate
  Other Names: Qsymia; Phentermine and topiramate
  Arms: VI-0521 Mid Dose (Phentermine 7.5 mg +Topiramate 46 mg); VI-0521 Top Dose (Phentermine 15 mg + Topiramate 92 mg)
Drug: Placebo oral capsule — Inactive drug
  Arms: Placebo
Behavioral: Lifestyle Modification — The lifestyle modification includes physical activity, behavior change, reduced calorie diet advice, and family support. This intervention is applied to all treatment groups.

SUMMARY:
This study is being conducted to assess weight loss efficacy, as determined by changes in body mass index (BMI), and safety of VI-0521 (Qsymia®) or placebo, taken for 56 weeks accompanied by a lifestyle modification program in obese adolescents age 12-16 years.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 12 years and < 17 years;
* BMI ≥ the 95th percentile, with documented history of failure to lose sufficient weight or failure to maintain weight loss in a lifestyle modification program;
* If female, must be using adequate contraception, defined as double barrier methods, stable hormonal contraception plus single barrier method, tubal ligation, or abstinence.

Exclusion Criteria:

* Type 1 diabetes;
* Congenital heart disease; clinically significant ECG abnormality;
* Clinically significant physical exam, vital signs, or laboratory abnormality; clinically significant hepatic or renal disease;
* Estimated Glomerular Filtration Rate (GFR; Schwartz formula) < 60 mL/minute;
* Clinically significant thyroid dysfunction as evidenced by signs, symptoms, or thyroid stimulating hormone (TSH) > 1.5 x Upper Limit of Normal;
* Obesity of known genetic or endocrine origin;
* History of bipolar disorder or psychosis, depression of moderate or greater severity, or presence or history of suicidal behavior or active suicidal ideation;
* Recent weight instability, or prior bariatric surgery;
* History of glaucoma or increased intraocular pressure;
* Current smoker or smoking cessation within 3 months of screening;
* Currently taking or plan on taking any of following medications during the study:

  * Anticonvulsants used for treatment of seizure disorder, including barbiturates, benzodiazepines, gamma-aminobutyric acid (GABA) analogues, hydantoins, phenyltriazines, succinimides, and other agents (valproic acid and its derivatives, carbamazepine and its derivatives, zonisamide, and felbamate);
  * Tricyclic antidepressants, monoamine oxidase inhibitors (MAOIs), lithium, levodopa, and dopamine receptor agonists;
  * Carbonic anhydrase inhibitors;
  * Insulin, Sulfonylureas (SFUs), glucagon-like peptide -1 (GLP-1) agonists, sodium glucose transporter-1 (SGLT-1), and SGLT-2 inhibitors;
  * Chronic systemic steroids (i.e. glucocorticoids, anabolic steroids) other than oral contraceptives;
  * Treatment for hyperactivity disorder; or
  * Over the counter, prescription medications, herbal agents and dietary supplements used with the intention to lose body weight.

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 223 (Actual)
Dates: Start 2019-05-02 (Actual); Primary Completion 2021-04-16 (Actual); Study Completion 2021-04-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Intend Research, LLC, Norman, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kelly AS, Bensignor MO, Hsia DS, Shoemaker AH, Shih W, Peterson C, Varghese ST. Phentermine/Topiramate for the Treatment of Adolescent Obesity. NEJM Evid. 2022 Jun;1(6):10.1056/evidoa2200014. doi: 10.1056/evidoa2200014. Epub 2022 Apr 30. PMID 36968652

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 26 study sites in the United States.
Pre-assignment Details: The study consisted of a Screening period of up to 28 days. Once confirmed participant meeting all study criteria, including laboratory values, participants were randomized to either placebo, Mid-dose, or Top-dose of VI-0521 (phentermine/topiramate [PHEN/TPM]), for a 56-week treatment period.
Groups:
- Placebo: Weeks 1-56: Placebo (Inactive drug) oral capsule, once daily; Weeks 1-56: Lifestyle Modification
- VI-0521 Mid Dose: Weeks 1-2: VI-0521 (PHEN/TPM 3.75 mg/23 mg) oral capsule, once daily; Weeks 3-56: VI-0521 (PHEN/TPM 7.5 mg/46 mg) oral capsule, once daily; Weeks 1-56: Lifestyle Modification
- VI-0521 Top Dose: Weeks 1-2: VI-0521 (PHEN/TPM 3.75 mg/23 mg) oral capsule, once daily; Weeks 3-12: VI-0521 (PHEN/TPM 7.5 mg/46 mg) oral capsule, once daily; Weeks 13-14: VI-0521 (PHEN/TPM 11.25 mg/69 mg) oral capsule, once daily; Weeks 15-56: VI-0521 (PHEN/TPM 15 mg/92 mg) oral capsule, once daily; Weeks 1-56: Lifestyle Modification
Period: Overall Study
Arm/Group | Placebo | VI-0521 Mid Dose | VI-0521 Top Dose
Started | 56 | 54 | 113
Completed | 29 | 37 | 73
Not Completed | 27 | 17 | 40
Not completed — Adverse Event | 1 | 1 | 2
Not completed — Lost to Follow-up | 13 | 9 | 20
Not completed — Lack of Efficacy | 2 | 0 | 1
Not completed — Protocol Non-Compliance | 0 | 0 | 1
Not completed — Withdrawal by Subject / Parent / Legal Guardian | 10 | 6 | 14
Not completed — All Other Personal Reasons | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | VI-0521 Mid Dose | VI-0521 Top Dose | Total
Number analyzed (Participants) | 56 | 54 | 113 | 223
Age, Continuous [Median (Full Range); unit: years] | 14.0 [12 to 16] | 14.1 [12 to 16] | 13.9 [12 to 16] | 14.0 [12 to 16]
Age, Customized [Count of Participants; unit: Participants]
  12-14 Years | 34 | 33 | 69 | 136
  15-16 Years | 22 | 21 | 44 | 87
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 28 | 63 | 121
  Male | 26 | 26 | 50 | 102
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 25 | 34 | 72
  Not Hispanic or Latino | 42 | 28 | 79 | 149
  Unknown or Not Reported | 1 | 1 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 42 | 36 | 71 | 149
  Black or African American | 10 | 14 | 36 | 60
  Other | 4 | 4 | 4 | 12
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 56 | 54 | 113 | 223
BMI Categories [Count of Participants; unit: Participants]
  ≥95th to <99th percentile | 26 | 23 | 33 | 82
  ≥99th percentile | 30 | 30 | 79 | 139
  Missing | 0 | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Mean % Change in Body Mass Index (BMI)
Description: Mean % change in BMI from Baseline to Week 56
Time Frame: Baseline to Week 56
Measure: Least Squares Mean (Standard Error); unit: Percentage Change
Arm/Group | Placebo | VI-0521 Mid Dose | VI-0521 Top Dose
Number analyzed (Participants) | 56 | 54 | 113
Percentage Change | 3.34 (1.441) | -4.78 (1.302) | -7.11 (1.011)
Statistical Analysis 1: Comparison: Placebo vs VI-0521 Mid Dose vs VI-0521 Top Dose; Test type: Superiority; p < 0.0001, Mixed Models Analysis

2. Secondary Outcome: Percentage of Subjects Achieving at Least 5% BMI Reduction at Week 56
Time Frame: Baseline to Week 56
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | VI-0521 Mid Dose | VI-0521 Top Dose
Number analyzed (Participants) | 56 | 54 | 113
percentage of participants | 13.6 | 44 | 52.2
Statistical Analysis 1: Comparison: Placebo vs VI-0521 Mid Dose vs VI-0521 Top Dose; Test type: Superiority; p < 0.0017, Cochran-Mantel-Haenszel

3. Secondary Outcome: Percentage of Subjects Achieving at Least 10% BMI Reduction at Week 56
Time Frame: Baseline to Week 56
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | VI-0521 Mid Dose | VI-0521 Top Dose
Number analyzed (Participants) | 56 | 54 | 113
percentage of participants | 4.5 | 33.5 | 44.4

4. Secondary Outcome: Percentage of Subjects Achieving at Least 15% BMI Reduction at Week 56
Time Frame: Baseline to Week 56
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | VI-0521 Mid Dose | VI-0521 Top Dose
Number analyzed (Participants) | 56 | 54 | 113
percentage of participants | 2.9 | 13.6 | 28.9

5. Secondary Outcome: Change in Waist Circumference at Week 56
Description: Change in waist circumference from Baseline to Week 56
Time Frame: Baseline, Week 56
Measure: Least Squares Mean (Standard Error); unit: Centimeter
Arm/Group | Placebo | VI-0521 Mid Dose | VI-0521 Top Dose
Number analyzed (Participants) | 56 | 54 | 113
Centimeter | 0.61 (1.397) | -5.03 (1.376) | -6.98 (1.072)

6. Secondary Outcome: Change in Whole Body Insulin Sensitivity Index (WBISI) (Matsuda) at Week 56
Description: Mean changes in glycemic parameters [Whole Body Insulin Sensitivity Index (WBISI) (Matsuda)] from baseline to Week 56. The Oral Glucose Tolerance Test (OGTT) were performed at Baseline and Week 56 using 75 g oral glucose load; blood samples were obtained at baseline and at 2 hours post glucose load for evaluation of both glucose and insulin levels. Insulin Sensitivity was measured by obtaining glucose and insulin levels in a fasting state and at 2 hours after administration of oral glucose load. Matsuda index = 10,000/SQRT [glucose concentration (mg/dL) (fasting)*insulin concentration (uIU/mL) (fasting)*glucose concentration (mg/dL) (2 hours after glucose load)*insulin concentration (uIU/mL) (2 hours after glucose load)], with higher numbers indicating better insulin sensitivity.
Time Frame: Baseline, Week 56
Population: The number of subjects with values at both time points (Baseline and Week 56)
Measure: Least Squares Mean (Standard Error); unit: Index
Arm/Group | Placebo | VI-0521 Mid Dose | VI-0521 Top Dose
Number analyzed (Participants) | 56 | 54 | 113
Index | -3.7 (8.887) | -3.93 (7.647) | -2.99 (6.445)

7. Secondary Outcome: Change in Fasting Insulin at Week 56
Description: Change in fasting insulin from Baseline to Week 56
Time Frame: Baseline, Week 56
Measure: Least Squares Mean (Standard Error); unit: uIU/mL
Arm/Group | Placebo | VI-0521 Mid Dose | VI-0521 Top Dose
Number analyzed (Participants) | 56 | 54 | 113
uIU/mL | -3.32 (8.956) | -11.47 (7.433) | -7.99 (6.299)

8. Secondary Outcome: Percent Change in Triglycerides From Baseline to Week 56
Time Frame: Baseline, Week 56
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Placebo | VI-0521 Mid Dose | VI-0521 Top Dose
Number analyzed (Participants) | 56 | 54 | 113
Percent Change | 5.56 (8.407) | -6.18 (7.958) | -5.59 (7.17)

9. Secondary Outcome: Percent Change in HDL-C From Baseline to Week 56
Time Frame: Baseline, Week 56
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Placebo | VI-0521 Mid Dose | VI-0521 Top Dose
Number analyzed (Participants) | 56 | 54 | 113
Percent Change | -4.3 (15.1) | 2.11 (11.501) | 0.65 (9.561)
Statistical Analysis 1: Comparison: Placebo vs VI-0521 Mid Dose vs VI-0521 Top Dose; Test type: Superiority; p = 0.7465, Mixed Models Analysis

10. Secondary Outcome: Change From Baseline in Systolic Blood Pressure at Week 56
Time Frame: Baseline, Week 56
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | VI-0521 Mid Dose (Phentermine 7.5 mg +Topiramate 46 mg) | VI-0521 Top Dose (Phentermine 15 mg + Topiramate 92 mg)
Number analyzed (Participants) | 56 | 54 | 113
mmHg | 2.86 (1.63) | 0.09 (1.503) | 1.84 (1.111)

11. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure at Week 56
Time Frame: Baseline, Week 56
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | VI-0521 Mid Dose (Phentermine 7.5 mg +Topiramate 46 mg) | VI-0521 Top Dose (Phentermine 15 mg + Topiramate 92 mg)
Number analyzed (Participants) | 56 | 54 | 113
mmHg | 3.41 (1.51) | 0.24 (1.322) | 1.22 (0.989)

ADVERSE EVENTS:
Time Frame: About 1 year (from the time when the subject provides written informed consent and extends until 28 calendar days after the last dose of the investigational product is administered).
Arm/Group | Placebo | VI-0521 Mid Dose | VI-0521 Top Dose
All-Cause Mortality (participants affected / at risk) | 0/56 | 0/54 | 0/113
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/54 | 2/113
Other Adverse Events (participants affected / at risk) | 20/56 | 11/54 | 18/113
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=56) | VI-0521 Mid Dose (N=54) | VI-0521 Top Dose (N=113)
Depression (Psychiatric disorders) | 0 | 0 | 1
Suicidal Ideation (Psychiatric disorders) | 0 | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=56) | VI-0521 Mid Dose (N=54) | VI-0521 Top Dose (N=113)
COVID-19 (Infections and infestations) | 4 | 2 | 4
Upper respiratory tract infection (Infections and infestations) | 4 | 1 | 4
Nasopharyngitis (Infections and infestations) | 3 | 1 | 2
Headache (Nervous system disorders) | 5 | 4 | 5
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-06-21): https://cdn.clinicaltrials.gov/large-docs/45/NCT03922945/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-01): https://cdn.clinicaltrials.gov/large-docs/45/NCT03922945/SAP_001.pdf